CLINICAL TRIAL: NCT03422263
Title: Early Performance in Patients With Type-II-Diabetes Mellitus Under New Treatment With SGLT-2-Inhibitors Compared to Control Groups.
Brief Title: Performance Under SGLT-2-Inhibitors in Humans
Acronym: PUSH
Status: Completed | Type: Observational
Sponsor: Berner Klinik Montana (Other)
Responsible Party: Principal Investigator, Devine Frundi, Lead physician of internal medicine (Leitender Arzt Medizin), Berner Klinik Montana
Other Study IDs: Bernerklinik
Record Dates: First submitted 2018-01-23; First posted 2018-02-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: SGLT-2-Inhibitor, Empagliflozin, Canagliflozin, Dapagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with T2DM under new therapy with SGLT-2-Inhibitors: Patients with T2DM under new therapy with SGLT-2-Inhibitors (Empagliflozin 10 mg per day, Dapagliflozin 10 mg per day, Canagliflozin 100 mg per day) at baseline.
- Patients with T2DM without SGLT-2-Inhibitors.: Patients with T2DM without therapy with SGLT-2-Inhibitors (Empagliflozin 10 mg per day, Dapagliflozin 10 mg per day, Canagliflozin 100 mg per day) at baseline.
- Patients without T2DM manifesting similar comorbidities: Patients without T2DM manifesting similar comorbidities (Haemoglobin value, renal function, similar body mass index, cardiovascular disease profile)

SUMMARY:
The PUSH Study is conceived to investigate the early effects of SGLT-2-Inhibitors on the physical performance of patients with Type-II-Diabetes mellitus compared to patients under other therapy regimes. Patients shall be divided into 3 groups: I - Patients with type II diabetes mellitus under new treatment with an SGLT2-Inhibitor. II - Patients with type II diabetes mellitus without SGLT-2- Inhibitor medication. III - Patients without type II diabetes mellitus but with similar comorbidities to the previous groups.

DETAILED DESCRIPTION:
SGLT-2-Inhibitors have been shown to improve cardiovascular outcomes in patients with type II diabetes mellitus. Present evidence shows this effect to be not directly related to better serum glucose levels because the effect was measurable within several days of initiation of the treatment.

In a prospective single-centre double-blinded comparative observational study, other aspects of the effect of SGLT-2-Inhibitors shall be analyzed from patient registry, particularly the physical performance of patients under new treatment with SGLT-2-Inhibitors. Patient consent will be sort for the analysis of clinical data during the duration of stay.

Patients included in the registry suitable for analysis shall be divided into 3 groups: I - Patients with type II diabetes mellitus under new treatment with an SGLT2-Inhibitor. II - Patients with type II diabetes mellitus without SGLT-2- Inhibitor medication. III - Patients without type II diabetes mellitus but with similar comorbidities to the previous groups.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* ambulatory patients

Exclusion Criteria:

* relevant limitations in movement

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ambulatory patients above the age of 40 who provide informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Distance | 28 days
  Change in distance covered in metres (m).
Rate of perceived exertion | 28 days
  Change in modified Borg Scale as subjective assessment of moderate intensity physical activity ( Range 0 - 10)
Saturation | 28 days
  Change in saturation after exertion, expressed in %
Heart rate after exertion | 28 days
  Change in heart rate after exertion, expressed as bpm
Maximum oxygen uptake | 28 days
  Change in predicted VO2 max using distance covered in 6 minute walk test as follows 4.948 0.023*Mean 6 MWD (meters)

SECONDARY OUTCOMES:
Muscle anatomy | 28 days
  Change in muscle architecture parameter (MAP) measured as the mid-thigh diameter of the medial vastus muscle using B-mode sonography in centimètres (cm).
Muscle physiology | 28 days
  Muscle strength measured as hand grip in Newton using a hand dynamometer in kg
Biochemical | 28 days
  change in routine laboratory parameter related to muscle status using measurements of creatinine kinase in serum, CK in U/l
Subjective Assessment | 28 days
  Change in fatigue using a Fatigue Score questionnaire (FSMC) as assessed by patient (Range 20 - 100).
Echocardiographic parameters (function) | 28 days
  Change in left ventricular function using doppler readings of LVOT: LVEF using Dusmenil Formula SV/LVEDV expressed in %.
Muscle anatomy (echogenicity) | 28 days
  Change in muscle architecture parameter (MAP) measured as the mid-thigh echogenicity of the lateral vastus muscle, using image J software, arbitary units (AU)
Biochemical (metabolic function) | 28 days
  change in routine laboratory parameter related to metabolic function: Uric acid in serum, expressed in micromol/l
Body constitution (BMI) | 28 days
  change in body mass index measured as weight/height x height expressed in kg/m2
Body constitution (Hip circumference) | 28 days
  change in hip circumference measured at the maximum posterior protrusion of the buttocks in cm
Body constitution (Muscle mass predicted I) | 28 days
  change in muscle mass predicted using the Baumgartner equation 0.2487(BM) + 0.0483(ST)-0.1584(GQUAD) +0.0732(HGS) +2.5843(SEX) + 5.8828 in kg
Body constitution (Muscle mass predicted II) | 28 days
  change in muscle mass predicted using the muscle thickness of the forearm (4.89xMT-Ulna(cm)xHeight(m)-9.15) in kg

OTHER OUTCOMES:
Echocardiographic parameters (GLS) | 28 days
  Change in left ventricular systolic function using global longitudinal strain Imaging: GLS expressed as GLS avg in minus %.
Biochemical (NTproBNP) | 28 days
  change in routine laboratory parameter related to cardiac function using measurements of NTproBNP in ng/l
Echocardiographic parameters (LVEDV) | 28 days
  Change in left ventricular structure using B-mode Imaging: LVEDV in mm
Echocardiographic parameters (LAVI) | 28 days
  Change in left atrial structure structure using Biplane method: LAVI in ml/m2
Echocardiographic parameters (LV Massindex) | 28 days
  Change in left ventricular structure using B-mode Imaging: LV Massindex in g/m2
Echocardiographic parameters (E/e' avg) | 28 days
  Change in left ventricular diastolic function using Mitral inflow E velocity as obtained by pulsed-wave (PW) Doppler expressed E/e' avg ratio

CONTACTS AND LOCATIONS:
Overall Officials: Devine S Frundi, MD, Principal Investigator — Berner Klinik Montana
Locations (1):
- Berner Klinik Montana, Crans-Montana, Valais, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Results of the study for academic purposes for trainees to get an academic degree within Switzerland.

REFERENCES:
- [Derived] Kettig E, Kistler-Fischbacher M, de Godoi Rezende Costa Molino C, Bischoff-Ferrari HA, Frundi DS. Association of magnesium and vitamin D status with grip strength and fatigue in older adults: a 4-week observational study of geriatric participants undergoing rehabilitation. Aging Clin Exp Res. 2023 Aug;35(8):1619-1629. doi: 10.1007/s40520-023-02450-7. Epub 2023 Jun 7. PMID 37285075
- [Derived] Frundi DS, Kettig E, Popp LL, Hoffman M, Dumartin M, Hughes M, Lamy E, Fru YJW, Bano A, Muka T, Wilhelm M. Physical performance and glycemic control under SGLT-2-inhibitors in patients with type 2 diabetes and established atherosclerotic cardiovascular diseases or high cardiovascular risk (PUSH): Design of a 4-week prospective observational study. Front Cardiovasc Med. 2022 Jul 22;9:907385. doi: 10.3389/fcvm.2022.907385. eCollection 2022. PMID 35935634